CLINICAL TRIAL: NCT03160157
Title: Prospective Randomized Controlled Trial Comparing the Outcomes of Laparoscopic Cholecystectomy vs. Robotic Cholecystectomy
Brief Title: Comparing the Outcomes of Laparoscopic Cholecystectomy vs. Robotic Cholecystectomy
Acronym: RCT
Status: Withdrawn | Type: Observational
Why Stopped: No enrollment
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Antonio Gangemi, Professor of Clinical Surgery, University of Illinois at Chicago
Other Study IDs: 2016-0790
Record Dates: First submitted 2017-05-16; First posted 2017-05-19 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Gallbladder Diseases
MeSH Terms: conditions — Gallbladder Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- laparoscopic surgical group: Patients suitable for elective cholecystectomy with minimally invasive approach will be consented and randomized into either the robotic or laparoscopic group and both the patient and the operating physician will be notified which technique will be performed. Patients will be randomized to a 1:1 ratio. In order to eliminate bias in randomization, the investigators will be using an online resource available at: https://www.randomizer.org.
  After randomization, the investigators will complete a chart review that will follow the patients for a total of 30 days. The patient participation will be limited to the consent discussion and potential sign off. There will be no other clinic visits in regards to this research.
- robotic surgical group: Patients suitable for elective cholecystectomy with minimally invasive approach will be consented and randomized into either the robotic or laparoscopic group and both the patient and the operating physician will be notified which technique will be performed. Patients will be randomized to a 1:1 ratio. In order to eliminate bias in randomization, the investigators will be using an online resource available at: https://www.randomizer.org.
  After randomization, the investigators will complete a chart review that will follow the patients for a total of 30 days. The patient participation will be limited to the consent discussion and potential sign off. There will be no other clinic visits in regards to this research.

SUMMARY:
This research is being done to examine which minimally invasive surgical approach is associated with the best outcomes when performing cholecystectomy surgery: laparoscopic or robotic?

Laparoscopic and robotic approaches are similar surgical procedures using small incisions. The laparoscopic approach is largely used for the removal of the gallbladder (cholecystectomy).

At UIC, the investigators perform the majority of the gallbladder surgeries through the robotic approach and only a few using the laparoscopic approach. The robotic surgical tools allows the surgeon the same freedom of movement as a human wrist, while using a 3D camera view.

The laparoscopic and robotic surgical approaches both represent minimally invasive surgery approach and are associated with less pain, faster recovery and better cosmetic outcomes when compared to traditional open surgery. It is not currently known which approach is better.

DETAILED DESCRIPTION:
Laparoscopic approach is largely used for cholecystectomy surgery. Here, at UIC, however the investigators perform many surgeries of the gallbladder through robotic approach.

However, the investigators do also perform this surgery using the laparoscopic approach at UIC. Laparoscopic and robotic surgery represent both minimally invasive approach and are associated with less pain, faster recovery and better cosmetic outcomes when compared to traditional open surgery. The majority of cholecystectomies in USA are still being done with laparoscopic approach though. However, the number of centers switching to the more technologically advanced robotic approach is growing exponentially.

A recent paper has been published indicating that the robotic approach may decrease the rate of open conversion (traditional, open abdomen surgery) in cholecystectomy operations in comparison to laparoscopic approach1. Open conversion implies removal of the minimally invasive instruments (straight for laparoscopy and robotic with Endowrist® feature) from the patient's abdominal cavity and the creation of a large incision that starts in the midline, 2-5 cm below the xiphoid bone, extending in parallel with the costal margin for about 20 cm and going toward the right flank.

There is sparse literature comparing outcomes of cholecystectomy between the laparoscopic and robotic approaches and no other major studies that focus on just this procedure.

The investigators have already investigated the outcomes of robotic gallbladder surgery vs. laparoscopic surgery and published these data in a retrospective study, however the investigators are unsure if a prospective study would yield similar results.

Specific Aim:

The investigators would like to start a prospective randomized study to achieve definitive scientific evidence that will help determine which minimally invasive surgical approach is associated with the best outcomes when performing the removal of the gallbladder (cholecystectomy): laparoscopic or robotic?

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Any of the pre-operative diagnoses including chronic cholecystitis, acute cholecystitis, benign neoplastic disease of the gallbladder or pre-cancerous conditions of the gallbladder (polyps, adenomyomatosis), symptomatic cholelithiasis, porcelain gallbladder and biliary dyskinesia.

Exclusion Criteria:

1. 17 years of age or younger
2. Patient's that do not consent
3. Patients in which cholecystectomy is not the primary procedure, patients undergoing single site laparoscopic or robotic cholecystectomy, pregnant females, and malignant neoplastic conditions of the gallbladder (e.g. adenocarcinoma).
4. Patients with robotic equipment unavailable at time of surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suitable for elective cholecystectomy with minimally invasive approach
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Determine which minimally invasive (small incisions) surgical approach is associated with the best outcomes when performing the removal of the gallbladder (cholecystectomy): laparoscopic or robotic? | 2 years
  The following outcome will be tracked: open conversion (was the patient converted to open surgical procedure for either of the minimally invasive procedures, yes or no?)
Determine which minimally invasive (small incisions) surgical approach is associated with the best outcomes when performing the removal of the gallbladder (cholecystectomy): laparoscopic or robotic? | 2 years
  The following outcome will be tracked: biliary injuries (Did the patient have biliary injuries? If so, what?)
Determine which minimally invasive (small incisions) surgical approach is associated with the best outcomes when performing the removal of the gallbladder (cholecystectomy): laparoscopic or robotic? | 2 years
  The following outcome will be tracked: biliary anomalies (did the patient have biliary anomalies? If so, what?)
Determine which minimally invasive (small incisions) surgical approach is associated with the best outcomes when performing the removal of the gallbladder (cholecystectomy): laparoscopic or robotic? | 2 years
  The following outcome will be tracked: blood loss did the patient have blood loss? If so, amount in ml?)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Gangemi, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Outpatient Care Center (OCC), Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Data will be coded and will be analyzed by the research staff only. No IPD will be shared with other researchers.

REFERENCES:
- [Background] Gangemi A, Danilkowicz R, Elli FE, Bianco F, Masrur M, Giulianotti PC. Could ICG-aided robotic cholecystectomy reduce the rate of open conversion reported with laparoscopic approach? A head to head comparison of the largest single institution studies. J Robot Surg. 2017 Mar;11(1):77-82. doi: 10.1007/s11701-016-0624-6. Epub 2016 Jul 19. PMID 27435700